CLINICAL TRIAL: NCT04588701
Title: Long Term Outcomes After Surgery for Anal Fistula
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Richard Burney, Professor Emeritus of Surgery, University of Michigan
Other Study IDs: HUM00168195
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Fistula in Ano
Keywords: anal fistula; fistulotomy; ano-rectal advancement flap; sphincter saving
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- persons with anal fistulas: all persons with anal fistulas treated by a single surgeon over 22 years
  Interventions: Procedure: surgical procedures commonly done for anal fistula

INTERVENTIONS:
Procedure: surgical procedures commonly done for anal fistula — Surgical procedures performed, including fistulotomy; fistulotomy with sphincter repair; seton; advancement flap; fistula plug;

SUMMARY:
Anal fistula is a common condition with a wide variety of clinical presentations, which can make evaluation and treatment challenging and surgical outcomes uncertain. This study was undertaken to identify lessons learned in the surgical treatment of 483 patients over a 20- year period leading to a pragmatic approach to treatment of this condition.

DETAILED DESCRIPTION:
The wide array of variations of anal fistulas makes them challenging both to classify and to treat. The aim of the study is to determine if a systematic approach to their evaluation and surgical treatment, regardless of how one wishes to classify them, can be based on careful assessment of sphincter length and of the anatomical and etiological characteristics of the fistula.

ELIGIBILITY:
Inclusion Criteria:

* anal fistulas

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all persons with anal fistulas treated by a single surgeon at the University of Michigan Hospital from January 1996 through December 2018
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 1996-01-11 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Number of patients who heal after simple or staged operations for fistula | typically 1 year, but up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Burney, MD, Principal Investigator — University of Michigan